CLINICAL TRIAL: NCT03814291
Title: A Dose Escalation Phase I Clinical Study to Evaluate the Tolerability and Safety of IBI302 in Patients With Wet Age-related Macular Degeneration (AMD)
Brief Title: A Dose Escalation Study of IBI302 in Patients With Wet Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI302A101
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — IBI302

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- cohort 1 IBI302 treated with first dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302
- cohort 2 IBI302 treated with second dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302
- cohort 3 IBI302 treated with third dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302
- cohort 4 IBI302 treated with fourth dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302
- cohort 5 IBI302 treated with fifth dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302
- cohort 6 IBI302 treated with sixth dose level of IBI302 (Experimental)
  Interventions: Drug: IBI302

INTERVENTIONS:
Drug: IBI302 — 0.05mg/eye;Intraocular injection
  Arms: cohort 1 IBI302 treated with first dose level of IBI302
Drug: IBI302 — 0.15mg/eye;Intraocular injection
  Arms: cohort 2 IBI302 treated with second dose level of IBI302
Drug: IBI302 — 0.5mg/eye;Intraocular injection
  Arms: cohort 3 IBI302 treated with third dose level of IBI302
Drug: IBI302 — 1mg/eye;Intraocular injection
  Arms: cohort 4 IBI302 treated with fourth dose level of IBI302
Drug: IBI302 — 2mg/eye;Intraocular injection
  Arms: cohort 5 IBI302 treated with fifth dose level of IBI302
Drug: IBI302 — 4mg/eye;Intraocular injection
  Arms: cohort 6 IBI302 treated with sixth dose level of IBI302

SUMMARY:
This study is designed for single-center, open-label, dose escalation phase I trial to evaluate the safety and tolerability of a single intravitreal injection of IBI302 in patients with wet AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 50 yrs. of age.
2. Active subfoveal CNV secondary to wet AMD, with lesion size ≤ 12 optic discs in the study eye.
3. BCVA score of 10-73 letters using ETDRS charts (in 4 meters) in the study eye.
4. Central macular sub-field thickness according to OCT of at least 250 micron.
5. Clear stereoscopic fundus photography is obtained while the lens or other media is clear.
6. Female subjects of childbearing age or male subjects with childbearing age female partner agree to take effective contraceptive measures from the screening period to 3 months after the end of treatment.
7. Willing and able to sign informed consent form and comply with visit and study procedures per protocol.

Exclusion Criteria:

1. Presence of other causes of CNV other than wet AMD in the study eye.
2. Presence of active diabetic retinopathy in the study eye.
3. Presence of uncontrolled glaucoma in the study eye (defined as IOP≥30mmHg despite the standardized treatment).
4. Prior retinal detachment in the study eye.
5. Prior any treatment of following in the study eye:

   1. Anti-VEGF therapy within 6 months prior to screening;
   2. Anti-complement therapy;
   3. Laser photocoagulation;
   4. Photodynamic therapy;
   5. Transpupillary thermotherapy
   6. Intraocular surgery;
   7. Intraocular or periocular glucocorticoid injection therapy within 6 months prior to enrollment;
6. Presence of any non-AMD disease that may affect visual acuity in the study eye
7. Prior anti-VEGF therapy within 1 month before study drug administration or plan of above anti-VEGF therapy in the non-study eye during the whole study.
8. Oral steroid drugs within 1 month before study drug administration.
9. Presence of active intraocular or periocular inflammation or infection.
10. Diabetic patients have any of the following conditions:

    1. Microvascular and macrovascular complications;
    2. HbA1c>7.5% when screening;
    3. Receiving more than two oral hypoglycemic agents;
    4. Receiving insulin or GLP-1 receptor agonist;
11. Hypertension (defined as systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg despite standard treatment);
12. Presence of any following laboratory abnormality:

    1. PLT<100×109/L, INR≥1.5ULN, APTT≥ 10 seconds more than ULN;
    2. ALT or AST >2ULN;
    3. Cr or Ur>1.5ULN;
13. Large or medium surgery, or unhealed surgical incisions, ulcers or fractures within 1 month before study drug administration.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Safety evaluation indicators | Baseline to Day43
  Decreasing of BCVA; b) Changes in intraocular pressure compared with baseline; c) Incidence, relatedness and severity of all adverse events, treatment emergent adverse events and serious adverse events;

SECONDARY OUTCOMES:
Efficacy evaluation indicators | Baseline to Day43
  Changes in central subfield thickness by OCT compared with baseline; b) Changes in CNV area by FA compared with baseline; c) Changes in BCVA compared with baseline.
Immunogenicity evaluation indicators | Baseline to Day43
  Positive rate of anti-drug antibody and neutralizing antibody
The area under the drug-time curve from 0 to time t (AUC0-t) | Baseline to Day43
The area under the curve at the time of 0-infinity (AUC0-∞) | Baseline to Day43
The peak concentration (Cmax) | Baseline to Day43
The peak time (Tmax) | Baseline to Day43
Clearance rate (CL) | Baseline to Day43
Half-life (t1/2) | Baseline to Day43
Free and total VEGF concentration | Baseline to Day43

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang S, Li T, Jia H, Gao M, Li Y, Wan X, Huang Z, Li M, Zhai Y, Li X, Yang X, Wang T, Liang J, Gu Q, Luo X, Qian L, Lu S, Liu J, Song Y, Wang F, Sun X, Yu D. Targeting C3b/C4b and VEGF with a bispecific fusion protein optimized for neovascular age-related macular degeneration therapy. Sci Transl Med. 2022 Jun;14(647):eabj2177. doi: 10.1126/scitranslmed.abj2177. Epub 2022 Jun 1. PMID 35648811